CLINICAL TRIAL: NCT03632655
Title: A Prospective, Randomized Trial Comparing Office-based MR-guided Prostate Biopsy Approaches: Transrectal Ultrasound-guided Biopsy Compared With a Transperineal Approach
Brief Title: A Prospective, Randomized Trial Comparing Office-based MR-guided Prostate Biopsy Approaches
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to procurement of new funding sources.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1705018187
Record Dates: First submitted 2018-08-09; First posted 2018-08-15 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer; Elevated PSA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Men will be randomized to receiving either TPM or TRUS targeted biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Transrectal Ultrasound Guided Biopsy (TRUS) (Active Comparator): Patients will receive a transrectal guided prostate biopsy
  Interventions: Procedure: prostate biopsy
- Transperineal Prostate Biopsy (Active Comparator): Patients will receive a transperineal prostate biopsy
  Interventions: Procedure: prostate biopsy

INTERVENTIONS:
Procedure: prostate biopsy — Men will be randomized to receiving either TPM or TRUS targeted biopsy

SUMMARY:
This randomized trial will compare the safety and efficacy of TPM versus TRUS biopsies performed in the outpatient setting. Primary endpoints will be pain as well as detection of clinically significant disease (defined as Gleason Score >=7 or cancer core length >=6 mm). Secondary endpoints will be detection of any prostate cancer, hospital re-admissions within 30 days, aborted procedures due to discomfort, procedure time, adverse events including hematuria, urinary retention, hematospermia, hematochezia, and infection, and patient-reported outcomes as measured on validated instruments such as International Prostate Symptom Scores (IPSS) and International Index of Erectile Function (IIEF-5). In men who subsequently elect to undergo radical prostatectomy for definitive treatment of their prostate cancer, Gleason scores at final pathology will be correlated to the Gleason scores obtained at time of biopsy.

DETAILED DESCRIPTION:
The feasibility of outpatient TPM has been well demonstrated.(Bianco & Martínez-Salamanca, 2016; Merrick et al., 2016; Smith et al., 2014) New technology now allows for fusion of MRI images with TPM devices, allowing for targeting of cancerous-appearing lesions on MRI. Such technology that fuses MRI-imaging with TRUS biopsy has become routine in U.S. clinical practice, with improved cancer detection rates as compared with standard TRUS.(Ahmed et al., 2017; Robertson, Emberton, & Moore, 2013)

This randomized trial will compare the safety and efficacy of TPM versus TRUS biopsies performed in the outpatient setting. Men will be randomized to receiving either TPM or TRUS targeted biopsy. All men will receive a urine culture within 2 weeks of biopsy and will be started on antibiotic prophylaxis prior to biopsy in accordance with AUA antimicrobial prophylaxis guidelines. Men with a positive urine culture will be treated with culture-specific antibiotics and must have a documented negative urine culture prior to biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Men 18 years or older with suspicion for prostate cancer based upon an elevated PSA, abnormal digital rectal examination, abnormal MRI
* Men on active surveillance with indication for biopsy

Exclusion Criteria:

* Men with active urinary tract infection, metastatic prostate cancer, history of colorectal surgery limiting insertion of transrectal probe, evidence of acute or chronic prostatitis, or concern for perineal cellulitis or fistula
* Men unfit to undergo prostate biopsy under local anesthesia
* Men with prior definitive therapy for prostate cancer, such as radiation therapy or partial gland ablation
* Men with contraindication to prostate MRI (claustrophobia, pacemaker, chronic kidney disease)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must have clinical suspicion of prostate cancer
Enrollment: 38 (Actual)
Dates: Start 2017-12-23 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Hu, M.D., M.P.H., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transrectal Ultrasound Guided Biopsy (TRUS) | Transperineal Prostate Biopsy
Started | 22 | 16
Completed | 0 | 0
Not Completed | 22 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transrectal Ultrasound Guided Biopsy (TRUS) | Transperineal Prostate Biopsy | Total
Number analyzed (Participants) | 22 | 16 | 38
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [59.5 to 70.5] | 69 [60 to 75.25] | 64 [60 to 74.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 22 | 16 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 9 | 21
  Unknown or Not Reported | 10 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 8 | 15
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 10 | 4 | 14
Region of Enrollment [Number; unit: participants]
  United States | 22 | 16 | 38

OUTCOME MEASURES:

1. Primary Outcome: Gleason Grade
Description: Detection of clinically significant disease
  Typical Gleason Scores range from 6-10. The higher the Gleason Score, the more likely that the cancer will grow and spread quickly.
  * Scores of 6 or less describe cancer cells that look similar to normal cells and suggest that the cancer is likely to grow slowly.
  * A score of 7 suggests and intermediate risk for aggressive cancer. Scoring a 7 means that the primary score (largest section of the tumor) scored a 3 or 4. Tumors with a primary score of 3 and a secondary score of 4 have a fairly good outlook, whereas cancers with a primary Gleason Score of 4 and a secondary score of 3, are more likely to grow and spread.
  * Scores of 8 or higher describe cancers that are likely to spread more rapidly, these cancers are often referred to as poorly differentiated or high grade.
Time Frame: 7 days post-biopsy
Population: The data was not collected due to the trial being terminated.
Arm/Group | Transrectal Ultrasound Guided Biopsy (TRUS) | Transperineal Prostate Biopsy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Patient-reported Pain, as Measured on a 0-10 Likert Scale
Description: Pain will be scored on a 0-10 Likert scale. 0 indicates no pain and high scores indicate greater pain.
Time Frame: At time of local anesthesia administration, initiation of biopsy, immediately following biopsy, 7 days post-biopsy, 3 months post-biopsy
Population: The data was not collected due to the trial being terminated.
Arm/Group | Transrectal Ultrasound Guided Biopsy (TRUS) | Transperineal Prostate Biopsy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Patient-reported Symptoms, as Measured by International Prostate Symptom Scores (IPSS) Questionnaire
Description: IPSS scores range from 1 to 35, with 1-7 indicating mild symptoms, 8-19 indicating moderate symptoms, 20-35 indicating severe symptoms.
Time Frame: baseline, 7 days post-biopsy, 30 days post-biopsy
Population: The data was not collected due to the trial being terminated.
Arm/Group | Transrectal Ultrasound Guided Biopsy (TRUS) | Transperineal Prostate Biopsy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Patient-reported Erectile Function, as Measured by International Index of Erectile Function (IIEF-5) Questionnaire
Description: IIEF-5 scores range from 1 to 25, with 1-7 indicating severe erectile dysfunction, 8-11 indicating moderate erectile dysfunction, 12-16 indicating mild-moderate erectile dysfunction, 17-21 indicating mild erectile dysfunction, and 22-25 indicating no erectile dysfunction.
Time Frame: baseline, 7 days post-biopsy, 30 days post-biopsy
Population: The data was not collected due to the trial being terminated.
Arm/Group | Transrectal Ultrasound Guided Biopsy (TRUS) | Transperineal Prostate Biopsy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Patient-reported Quality of Life, as Measured by EPIC-CP Questionnaire
Description: EPIC-CP comprises of 10 questions about the patient within the last four weeks.
  Questions 1,7,8,9 are each graded on a scale from 0-4 for a total of 12 points. Higher scores indicate worse quality of life with regards to urinary and sexual function.
  Questions 2-4 grade Urinary Incontinence Symptoms on a scale from 0-4 (max 12 points). Higher scores indicate worse urinary incontinence symptoms.
  Questions 5a-c grade Urinary Irritation/Obstructive Symptoms on a scale from 0-4 (max 12 poitns). Higher scores indicate worse urinary irritation/obstructive symptoms.
  Questions 6a-c grade Bowel Symptoms on a scale from 0-4 (max 12 points). Higher scores indicate worse bowel symptoms.
  Questions 10a-c grade Vitality/Hormonal Symptoms on a scale from 0-4 (max 12 points). Higher scores indicate worse vitality/hormonal symptoms.
  All scores are summed (max 60 points) to calculate the Overall Prostate Cancer QOL score. Higher score indicates worse patient-reported QOL.
Time Frame: baseline, 7 days post-biopsy, 30 days post-biopsy
Population: The data was not collected due to the trial being terminated.
Arm/Group | Transrectal Ultrasound Guided Biopsy (TRUS) | Transperineal Prostate Biopsy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Adverse Events
Description: Adverse events that have occurred, such as hospital re-admissions, aborted procedures due to discomfort, hematuria, urinary retention, hematospermia, hematochezia, and/or infection.
Time Frame: initiation of biopsy, immediately following biopsy, 7 days post-biopsy, 30 days post-biopsy
Population: The data was not collected due to the trial being terminated.
Arm/Group | Transrectal Ultrasound Guided Biopsy (TRUS) | Transperineal Prostate Biopsy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were not collected.
Description: Adverse event data were not collected due to the trial being terminated.
Arm/Group | Transrectal Ultrasound Guided Biopsy (TRUS) | Transperineal Prostate Biopsy
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Early termination due to procurement of new funding sources.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT03632655/Prot_SAP_000.pdf